CLINICAL TRIAL: NCT01874262
Title: A Study to Evaluate the Use of Mobile-phone Based Patient Support in Patients Diagnosed With Myocardial Infarction - SUPPORT
Brief Title: A Study to Evaluate the Use of Mobile-phone Based Patient Support in Patients Diagnosed With Myocardial Infarction
Acronym: SUPPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: ME-CV-1301
Record Dates: First submitted 2013-05-29; First posted 2013-06-11 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active group (Experimental): The software application used on the patients' smart phones in the active group, will contain both the e-diary and the mobile-phone based patient support. Patients will receive feedback by the mobile-phone based support not only on the data they enter into the mobile-phone based patient support but also on their reported daily ticagrelor use.
  Interventions: Device: Mobile-phone based patient support; Device: e-diary
- The control group (Placebo Comparator): In this group the patients will have access to the e-diary only, in which they will report their daily use of ticagrelor. The patients in the control group will not receive any feed-back.
  Interventions: Device: e-diary

INTERVENTIONS:
Device: Mobile-phone based patient support — The mobile-phone based patient support (investigational medical device) is a stand-alone software product used on the patients' own smart phone and used in addition to medical treatment.
  Arms: Active group
Device: e-diary — All patients (active and control group) participating in the study will report their daily use of ticagrelor in an e-diary which will be initiated on all study patients' smart phones.

SUMMARY:
The purpose of this study is to evaluate whether the mobile-phone based patient support has an impact on the adherence and persistence of ticagrelor treatment or on lifestyle changes that will have a positive impact on the cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written patient informed consent.
2. Patients must have a smart phone at their disposal and use it on a daily basis.
3. Female or male aged >18 years, diagnosed with a ST elevation Myocardial Infarction (STEMI) or non ST elevation Myocardial Infarction (NSTEMI) and treated with ticagrelor prior to inclusion into this study and for which the treating physician intend to continue prescribing ticagrelor according to the prescription recommendation.
4. Ability to read, understand and write Swedish.

Exclusion Criteria:

1. Participation in any clinical trial or device study in the last 30 days excluding prospective/retrospective register based studies that do not require any extra visits in addition to ordinary health care.
2. Patients not suitable for participation based on the investigators judgment for example:

   * Patients on treatment with triple antithrombotic treatment.
   * Patients on treatment with anticoagulantia.
   * Patients accepted/with a plan for thoracic surgery (CABG) or any other elective surgery that cannot be postponed until after study participation.
   * Patients with a life expectancy of less than 12 months.
   * Patients judged to be unable to follow a structured physical activity program.
3. Patients those are pregnant or lactating.
4. Patients involved in the planning and/or conduct of the study (applies to AstraZeneca staff and/or staff at the study site and application developer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Varenhorst, MD, PhD, Principal Investigator — Kardiologkliniken, Akademiska Sjukhuset Uppsala
Locations (13):
- Sweden (13):
  - Research Site, Gothenburg
  - Research Site, Jönköping
  - Research Site, Köping
  - Research Site, Linköping
  - Research Site, Nyköping
  - Research Site, Örebro
  - Research Site, Stockholm
  - Research Site, Sundsvall
  - Research Site, Umeå
  - Research Site, Uppsala
  - Research Site, Varberg
  - Research Site, Vaxjo
  - Research Site, Västerås

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled on 30 June 2013 and the last participant completed the study on 11 December 2014. Study participants were randomized from 15 centers in Sweden.
Pre-assignment Details: Before discharge from the hospital patients diagnosed with myocardial infarction and treated with ticagrelor were offered participation in the study and those that accepted and signed informed consent were randomized into one of the two study groups.
Groups:
- E-diary + Mobile-phone Based Patient Support: The software application used on the patients' smart phones in this group, contained both the e-diary and the mobile-phone based patient support. Patients received feedback by the mobile-phone based patient support not only on the data they entered into the mobile-phone based patient support but also on their reported daily ticagrelor use.
- E-diary: In this group the patients had access to the e-diary only, in which they reported their daily use of ticagrelor. Patients did not receive any feed-back except a reminder in case of a missing ticagrelor registration (which was applicable also for the other group receiving e-diary + the mobile-phone based patient support).
Period: Overall Study
Arm/Group | E-diary + Mobile-phone Based Patient Support | E-diary
Started | 91 | 83
Not Correctly Randomised | 2 | 0
Not Included Due to Tehnical Issues | 3 | 3
Completed | 86 | 80
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E-diary + Mobile-phone Based Patient Support | E-diary | Total
Number analyzed (Participants) | 86 | 80 | 166
Age, Customized [Mean (Standard Deviation); unit: years] | 56.8 (8.0) | 58.4 (8.6) | 57.5 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 71 | 63 | 134

OUTCOME MEASURES:

1. Primary Outcome: Non-adherence Score
Description: The primary composite endpoint was defined as a non-adherence score based on the combination of adherence failure events and treatment gaps. Adherence failure events were defined as 2 missed doses during an observation cycle of up to 7 days. The first registered missed dose of ticagrelor in the e-diary initiated an observation cycle of 1 week. If a second missed dose was registered during the week, this was considered an adherence failure event. The third missed dose initiated a new observation cycle, and the process restarted. If the second missed dose was registered after more than 1 week, this was not defined as an adherence failure event, but initiated a new observation cycle. Treatment gaps were defined as patient reported gaps of 4 consecutive doses.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Non-adherence score
Arm/Group | E-diary + Mobile-phone Based Patient Support | E-diary
Number analyzed (Participants) | 85 | 77
Non-adherence score | 16.6 (42.9) | 22.8 (41.3)
Statistical Analysis 1: Comparison: E-diary + Mobile-phone Based Patient Support vs E-diary; Test type: Superiority or Other; p = 0.025, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Only device related events were monitored in this study.
Arm/Group | E-diary + Mobile-phone Based Patient Support | E-diary
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An Investigator agrees to provide a copy of the publication to AstraZeneca (AZ) for review at least 60 days in advance of submission for publication. Investigators in multicenter (MC) studies agree to postpone MC publications until the earlier of the date of the first AZ-authorized MC publication or a period up to 18 months from study completion at all sites.